CLINICAL TRIAL: NCT02552160
Title: Non-interventional Study for Documentation of the Therapeutic Efficacy, Use and Tolerance of the Fixed-Dose Combinations (FDC) Duaklir® Genuair® (Aclidinium/Formoterol), Ultibro® Breezhaler® (Glycopyrronium/Indacaterol) and Anoro® (Umeclidinium/Vilanterol) in the Treatment of COPD Under Real Conditions in the Practices of Pneumologists, Internists, and General Practitioners
Brief Title: DETECT-Register DocumEnTation and Evaluation of a COPD Combination Therapy
Acronym: DETECT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D6570R00001
Record Dates: First submitted 2015-07-29; First posted 2015-09-17 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Fixed-dose Combination; LAMA/LABA (Long Acting Beta2-Agonists / Long Acting Muscarinic Antagonists); Inhaler; Aclidinium/Formoterol; Glycopyrronium/Indacaterol; Umeclidinium/Vilanterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients on Duaklir® Genuair®: Patients on fixed-dose combination Duaklir® Genuair® (Aclidinium/Formoterol)
- Patients on Ultibro® Breezhaler®: Patients on fixed-dose combination Ultibro® Breezhaler® (Glycopyrronium/Indacaterol)
- Patients on Anoro®: Patients on fixed-dose combination Anoro® (Umeclidinium/Vilanterol)

SUMMARY:
Prospective, multi-centre, non-interventional study to collect findings about the effects of LABA/LAMA (Long Acting Beta2-Agonists / Long Acting Muscarinic Antagonists) combination preparations on COPD (Chronic obstructive pulmonary disease) symptoms and quality of life under real conditions and to find out what types of patients are selected for this therapy by physicians.

DETAILED DESCRIPTION:
Retrospective aspect of documentation: For patients who have already been changed over to a fixed-dose combination, lung function parameters and CAT (COPD Assessment Test™) score from the time prior to the changeover will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Female/male of at least 40 years of age
* Patient diagnosed with COPD
* Patient was changed over within the last 3 months to a fixed-dose combination (FDC) (Aclidinium/Formeterol, Glycopyrronium/Indacaterol or Umeclidinium/Vilanterol), or there is already the intent to change the patient over to a fixed-dose combination (Aclidinium/Formeterol, Glycopyrronium/Indacaterol or Umeclidinium/Vilanterol).
* Lung function parameters and CAT score from the time prior to the changeover to an FDC are on record (within the last 6 months in the case of patients who have already been changed over) or are determined at the 1st visit (in the case of patients who have not yet been changed over but for whom such a changeover is intended).
* Signed declaration of consent

Exclusion Criteria:

* The prescribing information for the fixed-dose combinations (Duaklir® Genuair®, Ulibtro® Breezhaler® or Anoro®) list contraindications for the patient.
* Patient is pregnant, plans to become pregnant, or is nursing during the therapy period.
* Patient suffers from hypersensitivity to one of the active ingredients of the fixed-dose combinations.
* Patient is participating in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with COPD (Chronic obstructive pulmonary disease), who have been changed over within the last 3 months to one of the 3 listed fixed-dose combinations (FDC) or for whom such a changeover is intended, and whose lung function parameters and CAT (COPD Assessment Test™) score from the time prior to the changeover are available (within the last 6 months) or are determined at the time of the 1st visit, if this is planned as part of the routine treatment.
Sampling Method: Probability Sample
Enrollment: 3732 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Lung function | First visit (baseline)
  Assessment of FEV1 (Forced Expiratory Volume), FVC (Forced Vital Capacity)
Number of patients with concomitant diseases classified by diagnostic subgroups | First visit (baseline)
Number of patients receiving concomitant COPD (Chronic obstructive pulmonary disease) medication classified by therapeutic subgroups | First visit (baseline)
Number of patients with exacerbations within the previous 24 months | First visit (baseline)
  History of previous exacerbations that will be collected at first observational visit.

SECONDARY OUTCOMES:
Change in well-being and quality of life | First visit (baseline) to end of observational period at 12 months
  CAT (COPD Assessment Test™) questionnaire will be completed at each visit, approximately every 3 months.
Effect on the severity of the shortness of breath | First visit (baseline) to end of observational period at 12 months
  mMRC (modified Medical Research Council Dyspnea Scale) questionnaire will be completed at each visit, approximately every 3 months.
Change in the night-time and early-morning COPD symptoms | First visit (baseline) to end of observational period at 12 months
  NiSCI/EMSCI (Night-time symptoms of COPD Instrument / Early-morning symptoms of COPD instrument) questionnaire will be completed at each visit, approximately every 3 months.
Lung function | First visit (baseline) to end of observational period at 12 months
  Assessment of FEV1, FVC at each visit, approximately every 3 months.
Number of exacerbations by grade | First visit (baseline) to end of observational period at 12 months
  Number of exacerbations will be collected at each visit, approximately every 3 months
Adverse events | First visit (baseline) to end of observational period at 12 months
  Adverse events will be collected at each visit, approximately every 3 months.
Handling of inhaler | At 12 months
  Questionnaire regarding handling of inhaler by patient

CONTACTS AND LOCATIONS:
Locations (180):
- Germany (180):
  - Research Site, Aachen, D6570r00001
  - Research Site, Aldenhofen, D6570r00001
  - Research Site, Aldenhoven, D6570r00001
  - Research Site, Alzey, D6570r00001
  - Research Site, Ansbach, D6570r00001
  - Research Site, Apolda, D6570r00001
  - Research Site, Aschau, D6570r00001
  - Research Site, Auerbach, D6570r00001
  - Research Site, Augsburg, D6570r00001
  - Research Site, Bad Fallingbostel, D6570r00001
  - Research Site, Bad Hersfeld, D6570r00001
  - Research Site, Bad Honnef, D6570r00001
  - Research Site, Bad Lippspringe, D6570r00001
  - Research Site, Bad Reichenhall, D6570r00001
  - Research Site, Bad Sachsa, D6570r00001
  - Research Site, Bad Windsheim, D6570r00001
  - Research Site, Bad Wörishofen, D6570r00001
  - Research Site, Bamberg, D6570r00001
  - Research Site, Beelitz-Heilstätten, D6570r00001
  - Research Site, Bergisch Gladbach, D6570r00001
  - Research Site, Berlin, D6570r00001
  - Research Site, Biberach, D6570r00001
  - Research Site, Birkenwerder, D6570r00001
  - Research Site, Bitterfeld-Wolfen, D6570r00001
  - Research Site, Bochum, D6570r00001
  - Research Site, Bonn, D6570r00001
  - Research Site, Bottrop, D6570r00001
  - Research Site, Böhlen, D6570r00001
  - Research Site, Braunschweig, D6570r00001
  - Research Site, Bruchsal, D6570r00001
  - Research Site, Burghaslach, D6570r00001
  - Research Site, Burgwedel, D6570r00001
  - Research Site, Büchen, D6570r00001
  - Research Site, Celle, D6570r00001
  - Research Site, Chemnitz, D6570r00001
  - Research Site, Cologne, D6570r00001
  - Research Site, Cottbus, D6570r00001
  - Research Site, Darmstadt, D6570r00001
  - Research Site, Delitzsch, D6570r00001
  - Research Site, Dessau, D6570r00001
  - Research Site, Dorsten, D6570r00001
  - Research Site, Dortmund, D6570r00001
  - Research Site, Dresden, D6570r00001
  - Research Site, Duisburg, D6570r00001
  - Research Site, Düren, D6570r00001
  - Research Site, Düsseldorf, D6570r00001
  - Research Site, Eimsheim, D6570r00001
  - Research Site, Ellerstadt, D6570r00001
  - Research Site, Elsterwerda, D6570r00001
  - Research Site, Elterlein, D6570r00001
  - Research Site, Essen, D6570r00001
  - Research Site, Euerbach-Obbach, D6570r00001
  - Research Site, Euskirchen, D6570r00001
  - Research Site, Flensburg, D6570r00001
  - Research Site, Frankfurt, D6570r00001
  - Research Site, Frankfurt/M., D6570r00001
  - Research Site, Freiberg, D6570r00001
  - Research Site, Fürstenwalde, D6570r00001
  - Research Site, Fürth, D6570r00001
  - Research Site, Ganderkesee, D6570r00001
  - Research Site, Garching, D6570r00001
  - Research Site, Garmisch-Partenkirchen, D6570r00001
  - Research Site, Gauting, D6570r00001
  - Research Site, Gera, D6570r00001
  - Research Site, Gerwisch, D6570r00001
  - Research Site, Glienicke, D6570r00001
  - Research Site, Greiz, D6570r00001
  - Research Site, Gütersloh, D6570r00001
  - Research Site, Hagen, D6570r00001
  - Research Site, Halberstadt, D6570r00001
  - Research Site, Halle, D6570r00001
  - Research Site, Hamburg, D6570r00001
  - Research Site, Hanover, D6570r00001
  - Research Site, Hartenstein, D6570r00001
  - Research Site, Heidelberg, D6570r00001
  - Research Site, Hemmingen, D6570r00001
  - Research Site, Hettstedt, D6570r00001
  - Research Site, Hoyerswerda, D6570r00001
  - Research Site, Höchstadt an der Aisch, D6570r00001
  - Research Site, Ibbenbueren, D6570r00001
  - Research Site, Ingolstadt, D6570r00001
  - Research Site, Iserlohn, D6570r00001
  - Research Site, Issum, D6570r00001
  - Research Site, Jena, D6570r00001
  - Research Site, Karlsruhe, D6570r00001
  - Research Site, Kevelaer, D6570r00001
  - Research Site, Kleve, D6570r00001
  - Research Site, Koeln-Hoehenberg, D6570r00001
  - Research Site, Koeln-Rodenkirchen, D6570r00001
  - Research Site, Kolbermoor, D6570r00001
  - Research Site, Köthen, D6570r00001
  - Research Site, Krefeld, D6570r00001
  - Research Site, Kronach, D6570r00001
  - Research Site, Kyritz, D6570r00001
  - Research Site, Langenfeld, D6570r00001
  - Research Site, Leer, D6570r00001
  - Research Site, Leipzig, D6570r00001
  - Research Site, Leonberg, D6570r00001
  - Research Site, Lippstadt, D6570r00001
  - Research Site, Ludwigsburg-Ossweil, D6570r00001
  - Research Site, Ludwigshafen, D6570r00001
  - Research Site, Lübeck, D6570r00001
  - Research Site, Magdeburg, D6570r00001
  - Research Site, Mainz, D6570r00001
  - Research Site, Mannheim, D6570r00001
  - Research Site, Marburg, D6570r00001
  - Research Site, Markt Bibart, D6570r00001
  - Research Site, Menden, D6570r00001
  - Research Site, Merzig, D6570r00001
  - Research Site, Moers, D6570r00001
  - Research Site, Monheim, D6570r00001
  - Research Site, Mosbach, D6570r00001
  - Research Site, Mönchengladbach, D6570r00001
  - Research Site, Mühlhausen, D6570r00001
  - Research Site, München, D6570r00001
  - Research Site, Neumarkt, D6570r00001
  - Research Site, Neunkirchen, D6570r00001
  - Research Site, Neuruppin, D6570r00001
  - Research Site, Neusäß, D6570r00001
  - Research Site, Neustadt/Aisch, D6570r00001
  - Research Site, Neuwied, D6570r00001
  - Research Site, Nuremberg, D6570r00001
  - Research Site, Oettingen in Bayern, D6570r00001
  - Research Site, Oschatz, D6570r00001
  - Research Site, Oy-Mittelberg, D6570r00001
  - Research Site, Pirmasens, D6570r00001
  - Research Site, Potsdam, D6570r00001
  - Research Site, Pulheim-Braunweiler, D6570r00001
  - Research Site, Radebeul, D6570r00001
  - Research Site, Rastatt, D6570r00001
  - Research Site, Rathenow, D6570r00001
  - Research Site, Recklinghausen, D6570r00001
  - Research Site, Remscheid, D6570r00001
  - Research Site, Reutlingen, D6570r00001
  - Research Site, Rosenheim, D6570r00001
  - Research Site, Rostock, D6570r00001
  - Research Site, Roth, D6570r00001
  - Research Site, Rust, D6570r00001
  - Research Site, Rüdersdorf, D6570r00001
  - Research Site, Rüsselsheim am Main, D6570r00001
  - Research Site, Saalfeld, D6570r00001
  - Research Site, Saarbrücken, D6570r00001
  - Research Site, Saarlouis, D6570r00001
  - Research Site, Schleswig, D6570r00001
  - Research Site, Schmölln, D6570r00001
  - Research Site, Schönbrunn, D6570r00001
  - Research Site, Schwedt, D6570r00001
  - Research Site, Siegen, D6570r00001
  - Research Site, Simmern, D6570r00001
  - Research Site, Solingen, D6570r00001
  - Research Site, Sonsbeck, D6570r00001
  - Research Site, Spiesen, D6570r00001
  - Research Site, Spremberg, D6570r00001
  - Research Site, Steinhagen, D6570r00001
  - Research Site, Strausberg, D6570r00001
  - Research Site, Straßkirchen, D6570r00001
  - Research Site, Stuttgart, D6570r00001
  - Research Site, Sulzberg, D6570r00001
  - Research Site, Teterow, D6570r00001
  - Research Site, Teuchern, D6570r00001
  - Research Site, Thaleischweiler-Fröschen, D6570r00001
  - Research Site, Trier, D6570r00001
  - Research Site, Ulm, D6570r00001
  - Research Site, Unterwellenborn, D6570r00001
  - Research Site, Ursensollen, D6570r00001
  - Research Site, Voerde, D6570r00001
  - Research Site, Wallenhorst, D6570r00001
  - Research Site, Wardenburg, D6570r00001
  - Research Site, Waren, D6570r00001
  - Research Site, Warendorf, D6570r00001
  - Research Site, Wehrheim, D6570r00001
  - Research Site, Weilheim, D6570r00001
  - Research Site, Weißenburg, D6570r00001
  - Research Site, Weißwasser, D6570r00001
  - Research Site, Wiesbaden, D6570r00001
  - Research Site, Witten, D6570r00001
  - Research Site, Wittenberg, D6570r00001
  - Research Site, Worms, D6570r00001
  - Research Site, Wuppertal, D6570r00001
  - Research Site, Zwönitz, D6570r00001

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3934&filename=DETECT_Report_Synopsis_20180720_final_Redacted_f_CTgov.pdf